CLINICAL TRIAL: NCT00419965
Title: Measuring GRK2 in the Blood to Diagnose and Treat Patients With Heart Failure
Brief Title: Measuring G Protein-coupled Receptor Kinase-2 (GRK2) in the Blood to Diagnose and Treat Patients With Heart Failure
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Walter J. Koch PhD (PI), Thomas Jefferson University Office of Research Administration
Other Study IDs: 06C.358
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen serum/plasma - coded samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary objective of this study is to determine the utility of GRK2 to differentiate between normal patients and patient groups that differ by the presence/absence of HF symptoms, systolic or diastolic left ventricular dysfunction, and risk factors; and to evaluate if a new assay provides similar values as traditional methods for measuring GRK2 levels.

DETAILED DESCRIPTION:
This study seeks to define a beta-adrenergic receptor kinase molecule in the blood and its role as an improved biomarker to be used for the diagnosis, assessment and management of patients with heart failure. We will test blood cell samples for the levels of this molecule, called "G protein-coupled receptor kinase-2" (GRK2) using both the existing method of GRK2 quantification in the Koch laboratory and using a prototype enzyme immunoassay (EIA) method being developed by Johnson & Johnson, Ortho-Clinical Diagnostics (OCD).

ELIGIBILITY:
Inclusion Criteria:

* Normal Controls: Individuals without HF, hypertension, diabetes, hyperlipidemia, coronary artery disease or obesity;
* Group I: Symptomatic Subjects with Reduced LV Function, HF symptoms, EF ≤ 40%.
* Group II: Asymptomatic Patients with LV dysfunction, no HF symptoms (NYHA class I and ATS score 0 or 1, EF ≤ 40%.
* Group III: Symptomatic Subjects with Preserved LV Function, HF symptoms, EF ≥ 50%, and diastolic dysfunction.
* Group IV: Asymptomatic High Risk Subjects - Individuals with normal heart function, no HF symptoms (NYHA class I and ATS score 0 or 1), Preserved LV function (EF ≥ 50%), no diastolic dysfunction. Also possess one or more cardiovascular high risk factors: diagnosis of diabetes; hyperlipidemia; coronary artery disease; renal insufficiency; hypertension; age >70 years

Exclusion Criteria

* Pregnancy
* Not providing consent
* Inability to provide consent
* Participation in a clinical study involving an experimental therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population subjects includes individuals in a range of age groups with a diagnosis of heart failure or at least one cardiovascular risk factor along with a subset of normal control subjects.
Sampling Method: Probability Sample
Enrollment: 582 (Actual)
Dates: Start 2006-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter J. Koch, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States